CLINICAL TRIAL: NCT01355757
Title: Post-Operative Quality of Life Evaluation for Different Anesthesia Techniques for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Admir Hadzic, Dr., St. Luke's-Roosevelt Hospital Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-142
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Rotator Cuff Injury
Keywords: shoulder arthroscopy; 24-week follow-up; quality of life; rehabilitation achievement; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Baxter INFUSOR System (Experimental): Regional Analgesia INFUSOR system with Patient Control Module for post-operative analgesia
  Interventions: Drug: Single Injection of Local Anesthetic
- Single Injection of Local Anesthetic (Active Comparator): Single injection of 20 ml ropivacaine 0.5%
  Interventions: Device: Baxter INFUSOR System

INTERVENTIONS:
Device: Baxter INFUSOR System — Regional Analgesia INFUSOR system with Patient Control Module for post-operative analgesia
  Arms: Single Injection of Local Anesthetic
Drug: Single Injection of Local Anesthetic — Single injection of 20 ml ropivacaine 0.5%
  Arms: Baxter INFUSOR System

SUMMARY:
Randomized controlled trial on efficacy of single injection or continuous interscalene brachial plexus block on analgesia in patients having outpatient rotator cuff surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients who agree to participate in the study will be asked to sign the informed consent and the HIPAA form.

Inclusive criteria are:

* 18-75 years of age
* ASA physical status I-III
* BMI < 35 kg/m2

Exclusion Criteria:

* all open shoulder procedures
* patient having difficulty understanding the instruction on using the anesthetic infusion pump
* contraindications to administration of regional anesthesia (e.g., allergy to a local anesthetic, local infection and coagulopathy)
* significant neurologic disorders of the upper extremity
* psychiatric or cognitive disorders
* history of substance abuse or chronic opioid use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 24 weeks
  To describe rehabilitation achievement and quality of life during 24-week follow-up after shoulder arthroscopy and rotator cuff repair, and identify any association between type of anesthesia procedure and patients' quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Admir Hadzic, MD PhD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's-Roosevelt Hospital, New York, New York, United States